CLINICAL TRIAL: NCT06475326
Title: A Phase II Trial of Adebrelimab in Combination With NALIRIFOX for Conversion Therapy in Locally Advanced Pancreatic Cancer
Brief Title: Adebrelimab in Combination With NALIRIFOX in Locally Advanced Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xian-Jun Yu, Professor, Fudan University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CSPAC-29
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Oxaliplatin; irinotecan sucrosofate; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adebrelimab Combined with NALIRIFOX (Experimental): Adebrelimab: 20 mg/kg, intravenous infusion, administered on day 1, every four weeks as a cycle (Q4W)
  Chemotherapy:
  Oxaliplatin: 60mg/m2, intravenous infusion for 2 hours, administered on day 1 Irinotecan liposome: 50mg/m2, intravenous infusion for more than 90min, administered on the first day LV: 400mg/m2, intravenous infusion for 2 hours, administered on the first day 5-FU: 2400mg/m2, continuous intravenous infusion for 46h, every two weeks as a cycle (Q2W)
  Interventions: Drug: Adebrelimab; Drug: Oxaliplatin 100 MG; Drug: Irinotecan liposome; Drug: Calcium Folinate; Drug: Fluorouracil

INTERVENTIONS:
Drug: Adebrelimab — Adebrelimab ,20mg/Kg per time, Q4W
  Other Names: PD-L1
Drug: Oxaliplatin 100 MG — Oxaliplatin: 60mg/m2, Q2W
Drug: Irinotecan liposome — Irinotecan Liposome: 50mg/m2, Q2W
Drug: Calcium Folinate — Calcium Folinate: 400mg/m2, Q2W
  Other Names: LV
Drug: Fluorouracil — Fluorouracil: 2400mg/m2, Q2W

SUMMARY:
In this study, Adebrelimab combined with NALIRIFOX conversion therapy was performed in subjects with locally advanced pancreatic cancer to evaluate the efficacy and safety of conversion therapy with immunotherapy combined with chemotherapy, followed by different treatment methods such as surgery, continued conversion therapy, and advanced systemic therapy according to different transformation outcomes, to improve the survival benefit of subjects with locally advanced pancreatic cancer.

DETAILED DESCRIPTION:
In this study, Adebrelimab combined with NALIRIFOX conversion therapy was performed in subjects with locally advanced pancreatic cancer to evaluate the efficacy and safety of conversion therapy with immunotherapy combined with chemotherapy, followed by different treatment methods such as surgery, continued conversion therapy, and advanced systemic therapy according to different transformation outcomes, to improve the survival benefit of subjects with locally advanced pancreatic cancer.

To assess the surgical resection conversion rate of chemotherapy in addition to immunotherapy for unresectable locally advanced pancreatic cancer (LAPC).

To evaluate the changes in CA19-9 levels, objective response rate (ORR), R0/R1 resection rate, pathologic response (pCR/MPR), event-free survival (EFS), 1 year and 2 years and overall survival (1y-OS, 2y-OS, OS) before and after conversion therapy for unresectable locally advanced pancreatic cancer.

To assess perioperative safety (including surgical morbidity and mortality within 60 days). To evaluate the safety and tolerability of immunotherapy in combination with chemotherapy for conversion therapy for unresectable locally advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old;
2. Histologically or cytologically confirmed pancreatic ductal adenocarcinoma (preferably histologically confirmed);
3. Judged by the investigator to be unresectable locally advanced (unresectable criteria refer to the guidelines for the diagnosis and treatment of pancreatic cancer);
4. Total bilirubin ≤ 2 mg/dL (subjects with bile duct stents can be enrolled if bilirubin ≤ 2 mg/dL and no cholangitis after stent placement);
5. Have not received previous treatment for pancreatic cancer, including radiotherapy, chemotherapy, surgery, etc;
6. Have at least one measurable lesion (per RECIST 1.1 criteria). ECOG score is 0~1 points within 28 days before the first dose, laboratory tests with adequate organ function: Blood routine: WBC ≥3.0×109/L; ANC≥1.5×109/L；PLT≥100×109/L； HGB≥90 g/L; Liver function: AST≤2.5×ULN; ALT≤2.5×ULN； TBIL≤1.5×ULN; Renal function: Cr≤1.5×ULN or CrCl ≥60 mL/min; Coagulation function: INR≤1.5, APTT≤1.5×ULN ; There was no obvious abnormality in ECG.
7. Male subjects, as well as females of childbearing potential, must use contraception for 3 months from the start of the first dose to the last use of the study drug.

Exclusion Criteria:

1. Occurrence of distant metastases (for imaging suspicion of peritoneal cancer or ascites, histological or cytological verification such as laparoscopic exploration is required)
2. Medical history and complications: Subject has contraindications to surgical resection of pancreatic cancer; Subject has any known active autoimmune disease; Subject has any complications requiring systemic treatment with glucocorticoids such as prednisone (>10mg/day) or has used immunosuppressive drugs within 14 days prior to the first dose; Subject has received tumor vaccine or other immune-activating antitumor drugs (such as interferon, interleukin, thymosin or immune cell therapy) within 1 month before the first dose; Subjects are participating in other clinical trials or have received drug intervention from other clinical trials within 4 weeks prior to the first dose.; Subject has other malignancies requiring treatment; Subject has had a significant prior cardiovascular disease; Subject has a known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation
3. Laboratory tests: Subject tested positive for HIV serologically; Active hepatitis B (HbsAg positive and HBV-DNA ≥103copies/mL) or active hepatitis C (HCV antibody positive and HCV-DNA positive with the need for antiviral therapy).
4. Presence of allergies and adverse drug reactions: Presence of allergy or hypersensitivity to monoclonal antibodies; Presence of allergic reactions to leucovorin, 5-FU, irinotecan, oxaliplatin
5. Diseases or abnormal laboratory indicators that in the opinion of the investigator will affect the results of the study, or are not in the interest of the subjects, should be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Surgical Conversion Rate | 8 weeks
  The surgery is scheduled to take place after a minimum of 4 weeks from the last dose to allow the effects of the drug to wear off. The eligible subjects can undergo surgery within 8 weeks from the last dose.

SECONDARY OUTCOMES:
Pathologic response rate (pCR/MPR) | up to approximately 1 years
  pCR is defined as the proportion of subjects with complete disappearance of cancer cells from tumor lesions and lymph nodes. MPR is defined as the proportion of cancer cells in tumor lesions and lymph nodes < 10% of subjects, and the viable cells of carcinoma in situ are not included in the calculation of pCR. All tumor tissue and associated lymph node tissue samples should be grossly examined. Tissue samples should be sectioned at a thickness of 0.5 cm. Pathological evaluation should be performed for more extensive tumors with at least 1.0 cm thick sections.
Objective response rate (ORR) | up to approximately 1 years
  ORR=(CR+PR)/ITT*100%, and the binomial distribution was used to calculate its 95%CI.
Event-free survival (EFS) | up to approximately 1 years
  defined as the time from the start of treatment to the occurrence of any disease progression affecting surgery, postoperative disease progression or recurrence (per RECIST v1.1), or death due to any cause, whichever occurs first.
Overall survival (OS) | up to approximately 1 years
  defined as the time from the first dose to death from any cause, whichever occurs first. Participants who were still alive at the last follow-up had OS as data censored at the time of the last follow-up. For participants lost to follow-up, OS was counted as data censored as the time to last confirmed survival before loss-to-follow.

CONTACTS AND LOCATIONS:
Overall Officials: Weijing Zhang, Study Chair — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China